CLINICAL TRIAL: NCT03780595
Title: Efficacy and Safety of the Administration of the Passiflora Extract for Benzodiazepine Withdrawal in Institutionalized Older Adults: Clinical Trial Phase III
Brief Title: Passiflora Extract for Benzodiazepine Withdrawal
Acronym: SEDISTRESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutricion Medica S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SEDISTRESS
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Benzodiazepine Withdrawal (Disorder)
Keywords: Benzodiazepine; Withdrawal; passiflora

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passiflora (Experimental)
  Interventions: Drug: Passiflora incarnata
- Control (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Passiflora incarnata — Passiflora pills administration up to 6 pills per day
  Arms: Passiflora
Drug: Control — Control pills administration up to 6 pills per day
  Arms: Control

SUMMARY:
The aim of this clinical trials is compare the percentage of patient who achieve a reduction equal to or greater than 50% in the dose of benzodiazepines at 10 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 65 years old
2. Stable dose of benzodiazepines during last 3 months ( 4mg loracepam per day or equivalent)
3. Capable of giving consent and to answer the questionnaires according to researcher criteria

Exclusion Criteria:

1. Diagnosis of dementia moderate or severe (Test Minimental ≤ 20).
2. Acute confusional syndrome at the inclusion
3. Panic disorder
4. Obsesive-compulsive disorder
5. Any type of psycosis or bipolar disorder
6. Severe Parkison disease diagnosed
7. Current or past diagnosis of epilepsia
8. Recent stroke (last month)
9. Thyroid disorders not controlled or uncompensated
10. Alteration of deglutition
11. Previous drugs or alcohol abuse
12. Hospitalization (more than 24 hours) during the last month
13. Complex priority treatment (dialisis, chemotherapy...)
14. Life expectation less than 1 year
15. Benzodiazepines therapeutic uses not for anxiety or insomnio

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the percentage of patients who achieve to reduce the dose of benzodiazepines equal or more than 50% Reduction of the benzodiazepine dose | 10 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernando Agüera, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (8):
- Spain (8):
  - Residencia Albertia Moratalaz, Madrid
  - Residencia Amavir Ciudad Lineal, Madrid
  - Residencia Nogales Imperial, Madrid
  - Residencia Nogales Pontones, Madrid
  - Residencia Nogales Puerta de Hierro, Madrid
  - Residencia Albertia Valle de la Oliva, Majadahonda
  - Residencia Amavir San Agustín, San Agustín del Guadalix
  - Residencia Amavir Torrejón, Torrejón de Ardoz